CLINICAL TRIAL: NCT03911479
Title: Evaluation of Heart Rate Variability and Endothelial Function Three Months After Bariatric
Brief Title: Evaluation of Heart Rate Variability and Endothelial Function Three Months After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Eliete Bouskela (Unknown)
Responsible Party: Principal Investigator, Luiz Guilherme Kraemer-Aguiar, MD, MD, Rio de Janeiro State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRV_endo
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Short-term, non-blinded, non-randomized longitudinal study comparing obese patients undergoing bariatric surgery with those on clinical treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bariatric Surgery Group (Experimental)
  Interventions: Procedure: Bariatric Surgery
- Clinical Threatment (Other): Convencional treatment in a public tertiary outpatients care unit
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — Bariatric Surgery - convencionals Roux-en-Y gastric bypass (RYGB) and vertical gastrectomy (Sleeve; SG)

SUMMARY:
Was performed a longitudinal, study with twenty patients recruited for the bariatric surgery group and 20 for clinical treatment. The analysis of HRV and endothelial function were performed through peripheral arterial tonometry, in patients with obesity before and after three months of bariatric surgery. Were also analyzed GLP-1, insulin and glucose at fast, and 30 and 60 minutes. The results were compared in parallel with a control group with clinical treatment for obesity.

DETAILED DESCRIPTION:
To assess the pathophysiological mechanisms that leads the benefits in cardiovascular risk after bariatric surgery, through the autonomic nervous system and endothelial function, was performed a longitudinal, study with twenty patients recruited for the bariatric surgery group and 20 for clinical treatment.

The analysis of HRV and endothelial function were performed through peripheral arterial tonometry, in patients with obesity before and after three months of bariatric surgery.

Were also analyzed GLP-1, insulin and glucose at fast, and 30 and 60 minutes. The results were compared in parallel with a control group with clinical treatment for obesity.

ELIGIBILITY:
Inclusion Criteria:

Patients with obesity grade 3 [Body Mass Index (BMI) ≥ 40kg/m2] or grade 2 (BMI 35-39.9kg/m2) with comorbidities

Exclusion Criteria:

Current use of incretin mimetics or inhibitors of dipeptidyl peptidase-4 (DPP4); and history of a previous cardiovascular event (acute myocardial infarction, stroke or peripheral obstructive arterial disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-02-25 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Rate variability and endothelial function | 3 months
  assessed by peripheral arterial tonometry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomide Braga T, das Gracas Coelho de Souza M, Maranhao PA, Menezes M, Dellatorre-Teixeira L, Bouskela E, Le Roux CW, Kraemer-Aguiar LG. Evaluation of Heart Rate Variability and Endothelial Function 3 Months After Bariatric Surgery. Obes Surg. 2020 Jun;30(6):2450-2453. doi: 10.1007/s11695-020-04397-4. PMID 31916132